CLINICAL TRIAL: NCT06948162
Title: Exploration of the Utility of Dental-dedicated MRI for Dentistry
Status: Recruiting | Type: Observational
Sponsor: Donald Nixdorf (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry); Siemens Healthineers USA (Unknown)
Responsible Party: Sponsor-Investigator, Donald Nixdorf, Professor, University of Minnesota
Organization: University of Minnesota (Other)
Other Study IDs: University of Minnesota; Dentsply Sirona (Other: Dentsply Sirona)
Record Dates: First submitted 2025-03-28; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Dental Crowding; Dental Occlusion, Traumatic; Dental Pain; TMD/Orofacial Pain; TMD; Orthodontics; Endodontic Disease; Orthodontic Treatment
Keywords: Diagnosis; Magnetic resounance imaging
MeSH Terms: conditions — Crowding; Dental Occlusion, Traumatic; Toothache; Dental Pulp Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Dental patients: Dental patients receiving care that have imaging a part of routine care
  Interventions: Device: dental-dedicated MRI (ddMRI)

INTERVENTIONS:
Device: dental-dedicated MRI (ddMRI) — This descriptive observational research is comparative in design, that is comparing existing standard clinical dental images, not obtained in this study, to test (i.e., ddMRI) images.

SUMMARY:
This description observational research is comparative in design, that is comparing existing standard clinical dental images, not obtained in this study, to test (i.e., ddMRI) images. The standard clinical dental images consist of radiographs, such as bitewings, periapical, panoramic, cone-beam CT, and medical CT, as well medical MRIs of the temporomandibular joints (TMJ).The conceptualization of research questions, study designing, and interpretation of imaging data has and will involve content expertise in all ddMRI research.

DETAILED DESCRIPTION:
Patients recruited from dental clinics at the University of Minnesota School of Dentistry will be screened for eligibility and asked to complete an MRI safety screening questionnaire. Eligible individuals will be invited to participate in at least one study visit, during which an MRI scan will be performed. At the end of the session, participants will complete a short questionnaire about their experience during the scan.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Age: 18 years old or older
2. Receiving imaging for routine dental care
3. Does not have a serious medical condition
4. Is not pregnant or is not potentially pregnant
5. Is willing and able to give consent in English
6. Has the ability to manage their own calendar and schedule appointments
7. Willing to have a separate 2-hour appointment to have an MRI

Exclusion Criteria:

1. Unable to consent to participant in English
2. Serious health condition, which includes but not limited to renal failure/on dialysis, unstable heart disease (uncontrolled arrhythmia, cardiomyopathy and/or unable to lay flat, within 1 month of cardiac catheterization or myocardial infarction), unstable cerebral vascular disease (within 1 month of stroke and/or stent placement), diabetes (type I or II) not controlled by medication or diet, uncontrolled seizures, uncontrolled hyperthyroidism, non-allergic bronchospasm (chronic obstructive pulmonary disease and emphysema), uncontrolled movement disorder, and liver failure
3. Pregnant and/or intending to become pregnant,
4. Prisoner and/or not able to manage their own scheduling
5. Screen positive on MR safety questionnaire, specifically including people that have worked with or otherwise been exposure to metal particles and have the potential for such particles to be embed within them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental patients age 18 and older that are able to provide informed consent for themselves, being seen at the School of Dentistry at the UMN for routine dental care where diagnostic imaging is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Safety Assessment of ddMRI in Dental Patients | 1 year
  Evaluate the feasibility and safety of dental-dedicated MRI (ddMRI) in dental patients by assessing their experiences immediately following each scan. This will be done using an exit questionnaire designed to capture any sensations or discomforts that may have occurred during the scan. Participants will be asked to report the presence of various sensations, including but not limited to: nervousness, double vision, sleepiness, vertigo, lightheadedness, metallic taste, and feelings of warmth or cold. The collected responses will help determine the overall tolerability of ddMRI in this patient population.
Diagnostic Quality Assessment of ddMRI in Dental Patients | 1 year
  The diagnostic quality of dental-dedicated MRI (ddMRI) in dental patients will be evaluated through subjective ratings of its ability to identify various dentoalveolar anatomical structures. These ratings will be compared to those obtained from existing standard dental imaging modalities. Additionally, intra- and inter-rater reliability analyses will be conducted to assess the consistency of the ddMRI interpretations and their agreement with conventional dental imaging.
Anatomical landmark identification and inflammation detection | 3 years
  Compare the diagnostic efficacy of ddMRI versus existing clinical imaging (e.g., plain film, CT, MRI) in terms of identifying anatomical landmarks and detecting the presence of inflammation, as rated by dental specialist examiners.

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Nixdorf, DDS, MS, Principal Investigator — University of Minneosta; Laurance Gaalaas, DDS, MS, Study Director — University of Minneosta
Locations (1):
- Orofacial MRI Center at UMN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Orofacial Magnetic Resonance Imaging Center (OMRIC) facility at the UMN: a state-of-the-art research facility -1st in the nation- that supports oral and craniofacial imaging studies, particularly those involving MRI. — https://dentistry.umn.edu/omric